CLINICAL TRIAL: NCT04780841
Title: A Two-Part Proof-of-Concept Study: An Open-Label Dose-Ranging Phase (Part A) Followed by a Randomized, Single-Blind, Placebo-Controlled Phase (Part B) Evaluating the Safety and Efficacy of RDX013 for the Treatment of Hyperkalemia
Brief Title: A Study Evaluating the Safety and Efficacy of RDX013 for the Treatment of Hyperkalemia
Acronym: Redukx
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: RDX013-201
Record Dates: First submitted 2021-01-26; First posted 2021-03-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia

STUDY DESIGN:
Intervention Model Description: In Part A, treatment arms will be dosed based on the results from the previous arm. For Part B, one treatment arm from Part A will be selected
Who Masked: Participant
Masking Description: This is a two part study; Part A is open label and Part B is blinded to study participants (all drug labels for treatment arm and placebo will be identical)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- RDX013 Cohort 1 (Experimental): RDX013 low dose oral dosage, twice daily
  Interventions: Drug: RDX013
- RDX013 Cohort 2 (Experimental): RDX013 low, mid dose oral dosage, twice daily
  Interventions: Drug: RDX013
- RDX013 Cohort 3 (Experimental): RDX013 high, mid dose oral dosage, twice daily
  Interventions: Drug: RDX013
- RDX013 Cohort 4 (Experimental): RDX013 high dose oral dosage, twice daily
  Interventions: Drug: RDX013
- RDX013 Part B (Experimental): RDX013 dose from Part A oral dosage, twice daily
  Interventions: Drug: RDX013
- Placebo Part B (Placebo Comparator): oral dosage, twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RDX013 — RDX013 is an experimental drug that is a potassium secretagogue
  Arms: RDX013 Cohort 1; RDX013 Cohort 2; RDX013 Cohort 3; RDX013 Cohort 4; RDX013 Part B
Drug: Placebo — Placebo treatment that looks identical to experimental treatment
  Arms: Placebo Part B

SUMMARY:
The purpose of this study is to evaluate the ability of RDX013 to lower serum potassium in patients with chronic kidney disease with elevated serum potassium levels

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 to 85 years, inclusive
2. Serum potassium value 5.1 to <6.5 mmol/L
3. Chronic kidney disease with eGFR ≥20 to <60 mL/min/1.73m2
4. Able to understand and comply with the protocol
5. Willing and able to sign informed consent

Exclusion Criteria:

1. Pseudo-hyperkalemia signs and symptoms
2. Treatment with potassium-lowering drugs within 7 days prior to enrollment/randomization
3. Treatment with glucocorticoids
4. Uncontrolled Type 2 diabetes, defined as most recent historical HbA1c > 10%, or hospitalization to treat hyper- or hypo-glycemia in the past 3 months
5. Diabetic ketoacidosis
6. Severe heart failure, defined as NYHA (New York Heart Association) Class IV or hospitalization to treat heart failure in previous 3 months
7. History of bowel obstruction, severe gastrointestinal disorders, or major gastrointestinal surgery (e.g., large bowel resection)
8. Females who are pregnant, lactating, or not willing to use appropriate contraception

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Change in serum potassium; Part A | 1 week
  To evaluate the change of serum potassium from baseline to the end of treatment with different doses of RDX013 to identify the optimal dose for further evaluation in Part B of the study.
Change in serum potassium; Part B | 4 weeks
  To evaluate the difference between RDX013 and placebo in the change of serum potassium from baseline to the end of treatment.

SECONDARY OUTCOMES:
Exporatory Objective; time to serum potassium normalization | 4 weeks
  To evaluate the time to initial normalization of serum potassium level (≥3.5 to ≤5.0 mmol/L) during the initial 24 hours of treatment.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Horizon Research Group LLC, Coral Gables, Florida
  - Panax Clinical Research LLC, Miami Lakes, Florida
  - South Florida Research Phase I-IV; Inc., Miami Springs, Florida
  - NW Louisiana Nephrology Assoc, Shreveport, Louisiana
  - Clinical Research Consultants, Kansas City, Missouri
  - Mountain Kidney & Hypertension Associates, Asheville, North Carolina